CLINICAL TRIAL: NCT01955863
Title: Outpatient Radical Prostatectomy - Surgical and Anesthetic Considerations - Open Label Randomized Pilot Study
Brief Title: Outpatient Radical Prostatectomy - Surgical and Anesthetic Considerations
Acronym: ORP-SAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wesley Justino Magnabosco (Other)
Responsible Party: Sponsor-Investigator, Wesley Justino Magnabosco, member of urological team, Barretos Cancer Hospital
Organization: Barretos Cancer Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: OORP-2011
Record Dates: First submitted 2013-09-25; First posted 2013-10-08 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Prostatic Neoplasms
Keywords: Prostatic Neoplasms; Prostatectomy, Retropubic; Patient Discharge
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Patient Discharge

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- patient discharge on postoperative day 2 (Active Comparator): The patient was discharge on postoperative day 2 (as was done routinely)
  Interventions: Procedure: patient discharge on postoperative day 2
- patient discharge on postoperative day 1 (Experimental): The patient was discharge on postoperative day 1
  Interventions: Procedure: patient discharge on postoperative day 1
- patient discharge in the day of surgery (Experimental): The patient was discharge in the evening of the same day of surgery (average 12 hours of hospitalization)
  Interventions: Procedure: patient discharge in the day of surgery

INTERVENTIONS:
Procedure: patient discharge on postoperative day 2 — The patient was discharge on postoperative day 2 (as was done routinely)
  Arms: patient discharge on postoperative day 2
Procedure: patient discharge on postoperative day 1 — The patient was discharge on postoperative day 1
  Arms: patient discharge on postoperative day 1
Procedure: patient discharge in the day of surgery — The patient was discharge in the evening of the same day of surgery (average 12 hours of hospitalization)
  Arms: patient discharge in the day of surgery

SUMMARY:
Radical prostatectomy has become the gold standard treatment for prostate cancer.

Regarding of morbidity of access on open retropubic radical prostatectomy a lot of centers around the world start to develop laparoscopic and robotic approach over the past years. The problems regarding this techniques is that the pure laparoscopic prostatectomy shows a steep learning curve with a high initial complication rate, and the use of robotic assistance surgery despite of lower learning curve is associated with higher surgical supply and operative room costs. These costs may have a significant impact on overall cost of prostate cancer care especially in Brazil.

In Brazil, the open route for radical prostatectomy is still the most frequent approach. One of the disadvantages of open prostatectomy from the other surgeries is the longest hospital stay. However, the question of what length of stay after this operation is optimal and necessary is unresolved. In this trial the investigators have compared a randomized group of patients that had discharged on postoperative day 2, 1 and same day surgery. The investigators had intent to evaluate the feasibility of ambulatory open radical prostatectomy (patient discharge in the same day of surgery - average 12 hours of hospitalization) maintaining patient satisfaction and safety.

DETAILED DESCRIPTION:
Radical prostatectomy initially described by Walsh (1982) has become the gold standard treatment for prostate cancer and has evolved enormously over the last 25 years. Improvements include the use of smaller incisions, reduced blood loss, shorter hospital stays, and surgical refinement. Several large series with long-term follow-up have confirmed that this approach results in excellent cancer control and functional results in terms of preservation of erectile potency and urinary continence.

Regarding of morbidity of access on open retropubic radical prostatectomy a lot of centers around the world start to develop laparoscopic and robotic approach over the past years. The problems regarding this techniques is that the pure laparoscopic prostatectomy shows a steep learning curve with a high initial complication rate, and the use of robotic assistance surgery despite of lower learning curve is associated with higher surgical supply and operative room costs. These costs may have a significant impact on overall cost of prostate cancer care especially in Brazil where nowadays only have 3 centers with 5 robots.

In Brazil, the open route for radical prostatectomy is still the most frequent approach, mainly out of large cities. One of the disadvantages of open prostatectomy from minimally invasive surgeries is the longest hospital stay. However, the question of what length of stay after this operation is optimal and necessary is unresolved. In this trial the investigators have compared a randomized group of patients that had discharged on postoperative day 2, 1 and same day surgery. The investigators had intent to evaluate the feasibility of ambulatory open radical prostatectomy (patient discharge in the same day of surgery - average 12 hours of hospitalization) while maintaining patient satisfaction and safety.

ELIGIBILITY:
Inclusion Criteria:

* clinically localized Prostate Cancer (PCa)
* underwent open radical retropubic prostatectomy at Barretos' Cancer Hospital by a single primary surgeon (EFF)
* patients which the procedure went without any complications
* body mass index ≤ 30 kg/m2

Exclusion Criteria:

* Important comorbidities
* history of bleeding diathesis
* taking blood thinners

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-03; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of ambulatory open radical prostatectomy while maintaining patient satisfaction and safety. | 2 weeks postoperatively
  The endpoint regarding the survey is the comparison with standard group discharged at postoperative day 2. The satisfaction was considered non similar when there were more than 1 negative answer for any question or any patient in comparison to standard group in these questions: Do you consider your postoperative care adequate ? / Was your understanding of the necessary postoperative care adequate before enrolling for this study? Was your pain control adequate? / Was the length of hospitalization adequate? / Would you choose to have the procedure again with the same length of hospitalization? / Did you take any analgesic postoperatively after being discharged? / Did you take any analgesic postoperatively after being discharged? / Have you received adequate medical and nurse's care during the post-operative period? / Did you consider the access to the hospital easy if you needed it? / Would you recommend other men undergo this procedure the same way you?

CONTACTS AND LOCATIONS:
Overall Officials: Igor RM Franklin, MD, Principal Investigator — Barretos' Cancer Hospital; Eliney F Faria, PhD, Study Chair — Barretos' Cancer Hospital; Wesley J Magnabosco, MD, Study Director — Barretos' Cancer Hospital
Locations (1):
- Barretos' Cancer Hospital, Barretos, São Paulo, Brazil